CLINICAL TRIAL: NCT06264843
Title: Open, Prospective, Multicentre Study Addressing the Immediate Benefits and the Prognostic Value of Intraoperative Completion Control Following Infrainguinal Bypass Surgery in Chronic Limb-Threatening Ischemia (CLTI) Patients
Brief Title: Peripheral Bypass Trial for Completion Control
Acronym: PATENT
Status: Recruiting | Type: Observational
Sponsor: Medistim ASA (Industry)
Responsible Party: Sponsor
Other Study IDs: 724
Record Dates: First submitted 2024-02-09; First posted 2024-02-20 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Chronic Limb-Threatening Ischemia
Keywords: CLTI
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patency of lower extremity vein bypass grafts: Primary patency of lower extremity vein bypass grafts at one year
  Interventions: Device: MiraQ with Transit-Time Flow Measurement (TTFM) and L15 High Frequency Ultrasound (HFUS) probes

INTERVENTIONS:
Device: MiraQ with Transit-Time Flow Measurement (TTFM) and L15 High Frequency Ultrasound (HFUS) probes — Identify and validate intraoperative TTFM and HFUS findings (e.g. threshold values of Mean Graft Flow (MGF), MGF capacity, flow curve pattern, morphological issues)

SUMMARY:
The goal of the study is to identify and validate flow measurement and ultrasound images in patients undergoing vein bypass surgery below-knee and above ankle

ELIGIBILITY:
Inclusion Criteria:

* Chronic Limb-Threatening Ischemia as defined by presence of Peripheral Artery Disease (PAD) in combination with rest pain, gangrene, or a lower limb ulceration>2 weeks duration (ref Global Guidelines)
* Atherosclerotic infra-popliteal PAD
* Adequate distal anastomotic target (crural, tibial or popliteal below the knee with one single run-off) between knee and ankle distal to the stenotic/occluded segment.
* Available autogenous vein conduit based on preoperative vein mapping.
* Understand the nature of the procedure and willingness to comply with protocol. Attend follow-up appointments and provide written informed consent.

Exclusion Criteria:

* Bypass with artificial conduit or cryopreserved allografts
* Bypass for non-atherosclerotic lesions
* Life-expectancy less than 2 years
* Any psychological, developmental, physical or emotional disorder that the investigator believes would interfere with surgery or follow-up.
* Any condition that the investigator believes should exclude participation.
* Excessive risk for adverse events during open surgery as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic Limb-Threatening Ischemia patients scheduled to undergo a vein bypass with or without arterial inflow reconstruction to a below-knee and above ankle target
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Primary graft patency rate | at 1 year
  Freedom from any repeat graft intervention, graft thrombosis, or clinically significant stenosis (>70% by either Duplex criteria or angiographic imaging) in the bypass

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No